CLINICAL TRIAL: NCT00717587
Title: A Histopathologic and Imaging Study of Renal Cell Carcinoma Vasculature in the Setting of Sunitinib Therapy Prior to Cytoreductive Nephrectomy
Brief Title: Sunitinib Before and After Surgery in Treating Patients With Stage IV Kidney Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Keith T. Flaherty, Abramson Cancer Center of the University of Pennsylvania
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000600332; UPCC-10807; PFIZER-807184
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-01

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — motexafin gadolinium; Sunitinib; Comparative Genomic Hybridization; Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis; Immunohistochemistry; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: motexafin gadolinium
Drug: sunitinib malate
Genetic: comparative genomic hybridization
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymorphism analysis
Other: immunohistochemistry staining method
Other: iodine I-124 girentuximab
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sunitinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving it after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well sunitinib works when given before and after surgery in treating patients with stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To correlate histologic measures of tumor angiogenesis and VHL mutation/methylation status with clinical outcome in patients with stage IV renal cell carcinoma treated with sunitinib malate.
* To determine the effects of sunitinib malate on tumor vascular permeability by dynamic contrast-enhanced MRI and iodine I 124 chimeric monoclonal antibody G250 positron emission tomography (PET) after 2 weeks of therapy.
* To correlate steady-state plasma concentrations of sunitinib malate and angiogenic growth factors in serum with clinical outcome in these patients.

OUTLINE:

* Neoadjuvant therapy:Patients receive oral sunitinib malate once daily on days 1-14.
* Cytoreductive surgery: Patients undergo cytoreductive nephrectomy on day 16.
* Adjuvant therapy:Beginning at least 4 weeks after surgery, patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 42 days in the absence of disease progression or unacceptable toxicity.

Patients undergo dynamic contrast-enhanced MRI with motexafin gadolinium and positron emission tomography with iodine I 124 chimeric monoclonal antibody G250 at baseline and after completion of neoadjuvant sunitinib malate (prior to cytoreductive nephrectomy).

Patients undergo tumor tissue and blood sample collection periodically for correlative laboratory studies. Tumor tissue samples are analyzed for VHL mutations and other somatic genetic mutations by mutation analysis; allelic loss or gain by comparative genomic amplification; microvessel density (MVD) by immunohistochemical staining for CD34 and CD105; pERK, SMA, Ki-67, HIF-1α, CAIX, macrophage migration inhibition factor (MIF), and CREB by multicolor analysis; and VEGF-R1 and -R2 and other relevant antigen expression by validated assays. Blood samples are analyzed for pharmacokinetics; angiogenic growth factor levels (e.g., free VEGF, basic FGF, and other markers); and polymorphisms in VEGF, VEGFR, VHL, and HIF.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of renal cell carcinoma

  * AJCC stage IV disease
* Radiographic evidence of disease for which cytoreductive nephrectomy is deemed to be clinically indicated AND for which preoperative embolization is not deemed necessary by the surgeon
* No history or clinical evidence of brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,000/mm³
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Serum creatinine ≤ 2.0 times upper limit of normal (ULN) OR serum creatinine clearance ≥ 40 mL/min
* Total bilirubin ≤ 1.5 times ULN (< 3.0 times ULN in the presence of Gilbert's disease)
* AST/ALT ≤ 2.5 times ULN (≤ 5.0 times ULN in the presence of liver metastases)
* INR ≤ 1.5*
* PTT normal*
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pre-existing thyroid abnormality with thyroid-stimulating hormone that cannot be maintained in the normal range with medication
* No hypertension that cannot be controlled by medications (i.e., diastolic BP ≥ 100 mm Hg despite optimal medical therapy)
* No ongoing cardiac dysrhythmias ≥ grade 2 (according to NCI CTCAE v3.0)
* No other concurrent malignancies
* No concurrent serious illness including, but not limited to, any of the following:

  * Ongoing or active infection requiring parenteral antibiotics
  * Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, or unstable angina)
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Peripheral vascular disease ≥ grade 2 within the past year
  * Psychiatric illness/social situation that would limit compliance with study requirements NOTE: *Patients who are taking warfarin must have documentation of an INR ≤ 1.5 and PTT normal prior to the initiation of anticoagulation to rule out a baseline coagulopathy

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior radiotherapy and recovered
* Prior radiotherapy to a symptomatic site of metastatic disease is allowed
* No prior systemic therapy
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital), rifampin, or Hypericum perforatum (St. John's wort)
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Tumor regression as assessed by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Keith T. Flaherty, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States